CLINICAL TRIAL: NCT06215235
Title: Alleviation of Depressive Symptoms in People With Intellectual Disabilities
Brief Title: Implementation of Bright Light Therapy ID
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Margreet Vlastuin, Research Coordinator Quality, Erasmus Medical Center
Other Study IDs: Panama-10390; Wouters (Other: Erasmus MC)
Record Dates: First submitted 2023-09-08; First posted 2024-01-22 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Depressive Symptoms
Keywords: Depressive symptoms; Bright light therapy; Implementation; Intellectual disability
MeSH Terms: conditions — Depression; Intellectual Disability | interventions — Ultraviolet Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Persons involved in BLT: Persons with ID and staff who are involved in BLT. Either by receiving BLT, or by prescribing or facitating BLT.
  Interventions: Other: Bright light therapy

INTERVENTIONS:
Other: Bright light therapy — for 2 weeks the patient will take place for a 10.000lux lamp for 20-30 minutes.

SUMMARY:
Many adults with intellectual disabilities (ID) have depressive symptoms, which negatively impact their quality of life. A lot of of the non-medicinal forms of treatment are not or hardly suitable for people with ID. Bright light therapy (BLT) seems to be a good option. Earlier research has shown that BLT is applicable in this group and seems promising in terms of reducing depressive symptoms, without serious side effects.

In part 1 of this project we investigate the implementation of BLT at Amarant. We will take the lessons learned into part 2 of this project: the implementation of BLT at Abrona. We will evaluate this process and the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Involved in the implementation of BLT (staff) OR
* Involved in the prescription or application of BLT (staff/relatives) OR
* receiving BLT for their depressive symptoms (patients with ID)
* 18 years or older
* informed consent

Exclusion Criteria:

* n/a

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Patients are adult with an intellectual disability who have received BLT for their depressive symptoms.
  * Staff are adults (without ID) who work for one of the two care organizations and who are involved in the implementation or prescription or facilitation of BLT.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
acceptability | three times during study, 3-4 months in between
  Acceptability (Proctor et al., 2011) is the perception among implementation stakeholders that a given treatment, service, practice, or innovation is agreeable, palatable, or satisfactory. This will be measured by interviews.
appropriateness | three times during study, 3-4 months in between
  Appropriateness (Proctor et al., 2011) is the perceived fit, relevance, or compatibility of the innovation or evidence based practice for a given practice setting, provider, or consumer; and/or perceived fit of the innovation to address a particular issue or problem. This will be measured by interviews.
feasibility of the intervention | three times during study, 3-4 months in between
  Feasibility (Proctor et al., 2011) is defined as the extent to which a new treatment, or an innovation, can be successfully used or carried out within a given agency or setting. This will be measured by interviews.
fidelity | three times during study, 3-4 months in between
  Fidelity (Proctor et al., 2011) is defined as the degree to which an intervention was implemented as it was prescribed in the original protocol or as it was intended by the program developers. This will be measured by interviews and by case report study.
strategies | three times during study, 3-4 months in between
  Implementation strategies are methods to enhance the adoption, implementation and sustainability of a policy or intervention. This will be studied with interview data and logs.
Determinants | three times during study, 3-4 months in between
  Barriers and facilitators to BLT, measured by interviews using the Consolidated Framework for Implementation Research (CFIR, Damschroder et al., 2009)

SECONDARY OUTCOMES:
Depressive symptoms | 1 year
  Depressive symptoms measured by the Anxiety, Depression, and Mood Scale (ADAMS, Hermans et al., 2008). It contains 28 items, each can be scored 0 to 3. Minimum score 0 and maximum score 84 and higher scores mean worse outcome.
Behaviour | 1 year
  Behaviour that could be linked to depressive symptoms measured by the Aberrant Behaviour Checklist (ABC, Aman et al., 1985). It contains 58 items, each can be scored 0 to 3. Minimum score 0 and maximum score 174. Higher score means worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- ErasmusMC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided